CLINICAL TRIAL: NCT05027282
Title: A Prospective Study Evaluating the Safety and Effectiveness of the CLEAR + BRILLIANT TOUCH(R) Diode Laser 1440-nm and 1927-nm Combination Wavelength Treatment.
Brief Title: Safety and Effectiveness of the CLEAR + BRILLIANT TOUCH(R) Diode Laser 1440-nm and 1927-nm Combination Wavelength Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V01-CBT-401
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Photoaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm handpieces (Experimental)
  Interventions: Device: CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm handpieces.

INTERVENTIONS:
Device: CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm handpieces. — CLEAR + BRILLIANT TOUCH(R) diode laser 1440-nm and 1927-nm Combination Wavelength Treatment.

SUMMARY:
This is a prospective study of up to 30 subjects designed to assess the safety and effectiveness of a non-ablative fractional laser combination wavelength treatment for general resurfacing of photoaged skin. All study subjects will be treated on the whole face with the CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm handpieces. Subjects will be treated with a consecutive series of four (4) treatments spaced 1 month apart, along with follow-up study visits at one (1) and three (3) months after final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. 18 to 65 years of age.
3. Written and oral informed consent must be obtained.
4. No more than Mild (I) to Moderate (II) classification on Glogau Photodamage Scale.
5. Fitzpatrick skin types I-VI.
6. Fitzpatrick wrinkle & elastosis scale class I-II, score 1-6 (fine wrinkles and mild elastosis).
7. Ability to read, understand and sign the informed consent form.
8. Agree not to take any new medications (unless prescribed by the study investigator) or undergo any other procedures that may potentially treat photodamaged skin (any other aesthetic treatments) during the study.

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning to become pregnant during the study. 2 History of any type of allergic reaction to lidocaine. 3. Recent and/or active localized or systemic infections. 4. Diagnosis/possibility of actinic keratosis, melasma, rosacea, or other significant skin conditions (e.g. skin cancer, active infections, cold sores, open wounds, rashes, burns, inflammation eczema, psoriasis).

5. Predisposition to keloid formation or excessive scarring. 6. Diagnosis of a condition that may compromise the immune system, such as: HIV, lupus, scleroderma, and/or systemic infections.

7. Known sensitivity to light or photosensitizing agents/medications are being taken.

8. Systemic steroids (e.g. prednisone, dexamethasone), which should be rigorously avoided prior to and throughout course of the treatment.

9. Use of retinoids less than 2 weeks prior to or during the study to completion.

10. Individuals undergoing Accutane™ treatment or drugs in a similar class. 11. Having skin that is still recovering from a cosmetic procedure: such as a chemical peel, or mechanical peel, or laser resurfacing within the previous 6 months.

12. Having had Botox injections, neurotoxin injections, or dermal fillers (such as collagen) within the past four months.

13. Sunburn and/or recent sun exposure on the treatment area in the last 2 weeks.

14. Subjects must agree to seek the advice of their medical doctor regarding any known or suspicious skin condition before laser treatment.

15. Any condition or situation that would prevent the subject from safely completing all protocol requirements for participation.

16. Subjects who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Bhatt, Study Director — Bausch Health
Locations (1):
- Bausch Site 001, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm Handpieces
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm Handpieces
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Improvement in Photoaging Damage Appearance at 3 Months Post Treatment
Description: Improvement in the appearance of at least one measurement of photoaging damage (fine wrinkles, skin texture, dyschromia/pigment, skin radiance, pore size or overall appearance), each assessed by the investigator using the quartile improvement score comparing standard 2D baseline photograph captured via Canfield VISIA CA system. The Quartile Improvement Score ranges from 0 to 4, with 0 = 0%, 1 = 1% to 25%, 2 = 26% to 50%, 3 = 51% to 75%, and 4 = 76% to 100% improvement. Higher scores indicated greater improvement.
Time Frame: 3 months post treatment, up to 7 months
Population: Participants with 3 months of follow up were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm Handpieces
Number analyzed (Participants) | 26
units on a scale | 2.81 (0.9)

2. Secondary Outcome: Mean Improvement in Photoaging Damage Appearance at 1 Month Post Treatment
Description: as for outcome 1
Time Frame: 1 month post treatment, up to 5 months
Population: Participants with 1 month of follow up were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm Handpieces
Number analyzed (Participants) | 27
units on a scale | 2.59 (0.8)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | CLEAR + BRILLIANT TOUCH(R) 1440-nm and 1927-nm Handpieces
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT05027282/Prot_SAP_000.pdf